CLINICAL TRIAL: NCT00276094
Title: Efficacy and Safety of Ospemifene in the Treatment of Vulvar and Vaginal Atrophy (VVA) in Postmenopausal Women: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing Oral Ospemifene 30 and 60 Mg Daily Doses With Placebo
Brief Title: A Clinical Study to Evaluate Ospemifene in the Treatment of Vulvar and Vaginal Atrophy in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Collaborators: Hormos Medical (Industry); QuatRx Pharmaceuticals (Industry)
Responsible Party: Shionogi Clinical Trials Administrator, Shionogi
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-50310
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-03

CONDITIONS: Atrophy; Vaginal Diseases
Keywords: Urogenital atrophy; Vaginal atrophy; Vulvar and vaginal atrophy in postmenopausal women; Menopausal symptoms
MeSH Terms: conditions — Atrophy; Vaginal Diseases | interventions — Ospemifene

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Ospemifene 30 mg/day and nonhormonal vaginal lubricant (Experimental): Subjects will receive a single dose (1 tablet) of ospemifene 30 mg each morning with food for 12 weeks. The vaginal lubricant (K-Y® Brand Jelly) should be applied as needed and its use should be recorded in the medication diary. The first dose of the study drug will be administered at the clinic at Visit 2.
  Interventions: Drug: Ospemifene 30 mg; Drug: Nonhormonal vaginal lubricant
- Ospemifene 60 mg/day and nonhormonal vaginal lubricant (Experimental): Subjects will receive a single dose (1 tablet) of ospemifene 60 mg each morning with food for 12 weeks. The vaginal lubricant (K-Y® Brand Jelly) should be applied as needed and its use should be recorded in the medication diary. The first dose of the study drug will be administered at the clinic at Visit 2.
  Interventions: Drug: Ospemifene 60 mg; Drug: Nonhormonal vaginal lubricant
- Placebo tablets and nonhormonal vaginal lubricant (Placebo Comparator): Subjects will receive a single dose (1 tablet) of placebo each morning with food for 12 weeks. The vaginal lubricant (K-Y® Brand Jelly) should be applied as needed and its use should be recorded in the medication diary. The first dose of the study drug will be administered at the clinic at Visit 2.
  Interventions: Drug: Placebo; Drug: Nonhormonal vaginal lubricant

INTERVENTIONS:
Drug: Ospemifene 30 mg — 1 tablet (dose 30 mg/day) taken each morning with food for 12 weeks - from Visit 2 (Randomization, Day 1) to Visit 4 (Week 12).
  Arms: Ospemifene 30 mg/day and nonhormonal vaginal lubricant
Drug: Ospemifene 60 mg — 1 tablet (dose 60 mg/day) taken each morning with food for 12 weeks - from Visit 2 (Randomization, Day 1) to Visit 4 (Week 12).
  Arms: Ospemifene 60 mg/day and nonhormonal vaginal lubricant
Drug: Placebo — 1 tablet taken each morning with food for 12 weeks - from Visit 2 (Randomization, Day 1) to Visit 4 (Week 12).
  Arms: Placebo tablets and nonhormonal vaginal lubricant
Drug: Nonhormonal vaginal lubricant — Subjects should apply the vaginal lubricant as needed and record the usage in the medication diary.
  Other Names: K-Y® Brand Jelly

SUMMARY:
The purpose of this study is to determine whether ospemifene is more effective than placebo in the treatment of vulvar and vaginal atrophy (VVA) in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Naturally or surgically postmenopausal
* Moderate or severe symptoms of vaginal atrophy (ie, vaginal dryness, irritation or itching, difficult or painful urination, pain or bleeding with intercourse)
* Vaginal pH greater than 5.0
* 5% or fewer superficial cells in maturation index of vaginal smear

Exclusion Criteria:

* Evidence of endometrial hyperplasia, endometrial cancer, or other abnormal endometrial pathology
* Abnormal Pap smear
* Uterine bleeding of unknown origin or uterine polyps
* Current vaginal infection requiring medication

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 826 (Actual)
Dates: Start 2006-01; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi

RESULTS

PARTICIPANT FLOW:
Groups:
- Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant: Subjects received a single dose (1 tablet) of ospemifene 30 mg each morning with food for 12 weeks. The vaginal lubricant (K-Y® Brand Jelly) was applied as needed and its use was recorded in the medication diary. The first dose of the study drug was administered at the clinic at Visit 2.
- Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant: Subjects received a single dose (1 tablet) of ospemifene 60 mg each morning with food for 12 weeks. The vaginal lubricant (K-Y® Brand Jelly) was applied as needed and its use was recorded in the medication diary. The first dose of the study drug was administered at the clinic at Visit 2.
- Placebo Tablets and Nonhormonal Vaginal Lubricant: Subjects received a single dose (1 tablet) of placebo each morning with food for 12 weeks. The vaginal lubricant (K-Y® Brand Jelly) was applied as needed and its use was recorded in the medication diary. The first dose of the study drug was administered at the clinic at Visit 2.
Period: Overall Study
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Started | 282 | 276 | 268
Completed | 225 | 234 | 230
Not Completed | 57 | 42 | 38
Not completed — Adverse Event | 15 | 13 | 11
Not completed — Withdrawal by Subject | 14 | 14 | 12
Not completed — Protocol Violation | 16 | 7 | 10
Not completed — Lost to Follow-up | 8 | 6 | 4
Not completed — Other-Subject moved out of country | 1 | 0 | 0
Not completed — Other-Scheduled gastroplasty | 1 | 0 | 0
Not completed — Other-Lack of efficacy | 1 | 0 | 0
Not completed — Other-Refused follow-up visit | 1 | 0 | 0
Not completed — Other-Repeat safety labs-exclusionary | 0 | 1 | 0
Not completed — Other-Relocation | 0 | 1 | 0
Not completed — Other-Study medication lost | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant | Total
Number analyzed (Participants) | 282 | 276 | 268 | 826
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (6.27) | 58.6 (6.34) | 58.9 (6.09) | 58.6 (6.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 276 | 268 | 826
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Total number of participants in each arm/group do not match the "Overall Number of Baseline participants" in each Arm/group because "Race" and "Ethnicity" parameters have been combined to ensure faithful reproduction of each parameter, as mentioned in the CSR.
  Participants
    American Indian or Alaska Native | 0 | 2 | 1 | 3
    Asian | 5 | 4 | 6 | 15
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    Black or African American | 18 | 18 | 14 | 50
    White | 253 | 249 | 242 | 744
    Other | 6 | 2 | 4 | 12
    Missing value | 0 | 0 | 1 | 1
    Hispanic or Latino | 17 | 20 | 24 | 61
    Not Hispanic or Latino | 265 | 256 | 244 | 765
Height [Mean (Standard Deviation); unit: cm] | 161.9 (6.60) | 162.1 (6.42) | 162.3 (6.87) | 162.1 (6.62)
Weight [Mean (Standard Deviation); unit: kg] | 69.2 (13.06) | 68.4 (12.08) | 69.0 (12.90) | 68.9 (12.68)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.4 (4.51) | 26.0 (4.44) | 26.1 (4.37) | 26.2 (4.43)
Intact Uterus? [Number; unit: Participants]
  Yes | 129 | 128 | 122 | 379
  No | 153 | 148 | 146 | 447
Intact Cervix? [Number; unit: Participants]
  Yes | 133 | 133 | 129 | 395
  No | 149 | 143 | 139 | 431
Number (No.) of Pregnancies [Mean (Standard Deviation); unit: Pregnancies per participant] | 2.61 (1.834) | 2.39 (1.638) | 2.38 (1.525) | 2.46 (1.675)
No. of Vaginal Births [Mean (Standard Deviation); unit: Vaginal births per participant] | 1.78 (1.565) | 1.65 (1.478) | 1.59 (1.386) | 1.68 (1.480)
No. of Urinary Tract Infections in Past 6 Months [Number; unit: Participants]
  Missing values | 0 | 1 | 0 | 1
  0 | 247 | 239 | 242 | 728
  1 | 27 | 24 | 17 | 68
  2 | 7 | 9 | 8 | 24
  3 | 0 | 2 | 1 | 3
  4 or more | 1 | 1 | 0 | 2
Currently Experiencing Hot Flashes? [Number; unit: Participants]
  No | 110 | 102 | 113 | 325
  Yes | 172 | 174 | 155 | 501
No. of Days with Hot Flashes (/month) [Mean (Standard Deviation); unit: Days] | 19.7 (11.68) | 19.6 (11.49) | 19.6 (11.09) | 19.6 (11.41)
Previous Hormone Treatment [Number; unit: Partcipants]
  No | 232 | 222 | 218 | 672
  Yes | 50 | 54 | 50 | 154
Percentage of Parabasal Cells at Screening [Mean (Standard Deviation); unit: Percentage of Parabasal Cells] | 40.1 (38.33) | 39.3 (38.98) | 38.5 (37.60) | 39.3 (38.28)
Percentage of Superficial Cells at Screening [Mean (Standard Deviation); unit: Percentage of Superficial Cells] | 1.25 (2.907) | 1.04 (3.368) | 0.91 (2.635) | 1.07 (2.989)
Vaginal pH at Screening [Mean (Standard Deviation); unit: Vaginal pH] | 6.35 (0.736) | 6.37 (0.763) | 6.34 (0.732) | 6.35 (0.743)
Most Bothersome Vulvar and Vaginal Atrophy (VVA) Symptom (MBS) by Severity (Overall [Composite]) [Number; unit: Participants]
  None | 4 | 5 | 3 | 12
  Mild | 8 | 11 | 5 | 24
  Moderate | 121 | 109 | 121 | 351
  Severe | 148 | 150 | 136 | 434
MBS-Vaginal Dryness at Randomization [Number; unit: Participants] — Vaginal Dryness was assessed in 102, 118, and 104 subjects in the Ospemifene 30 mg, Ospemifene 60 mg, and Placebo groups, respectively.
  Participants
    Mild | 3 | 4 | 1 | 8
    Moderate | 47 | 61 | 62 | 170
    Severe | 52 | 53 | 41 | 146
MBS-Vaginal Pain with Sexual Activity at Randomization [Number; unit: Participants] — Vaginal Pain with Sexual Activity was assessed in 136, 120, and 122 subjects in the Ospemifeme 30 mg, Ospemifene 60 mg, and Placebo groups, respectively.
  Participants
    None | 3 | 4 | 2 | 9
    Mild | 3 | 3 | 1 | 7
    Moderate | 46 | 29 | 33 | 108
    Severe | 84 | 84 | 86 | 254
MBS-Vaginal and/or Vulvar Irritation or Itching at Randomization [Number; unit: Participants] — Vaginal and/or Vulvar Irritation or Itching was assessed in 39, 30, and 37 subjects in the Ospemifene 30 mg, Ospemifene 60 mg, and Placebo groups, respectively.
  Participants
    None | 1 | 0 | 1 | 2
    Mild | 2 | 4 | 3 | 9
    Moderate | 25 | 17 | 24 | 66
    Severe | 11 | 9 | 9 | 29
MBS-Difficult/Painful Urination at Randomization [Number; unit: Participants] — Difficult/Painful Urination was assessed in 3, 2, and 2 subjects in the Ospemifene 30 mg, Ospemifene 60 mg, and Placebo groups, respectively.
  Participants
    Moderate | 2 | 1 | 2 | 5
    Severe | 1 | 1 | 0 | 2
MBS-Vaginal Bleeding with Sexual Activity at Randomization [Number; unit: Participants] — Vaginal Bleeding with Sexual Activity was assessed in 1, 5, and 0 subjects in the Ospemifene 30 mg, Ospemifene 60 mg, and Placebo groups, respectively.
  Participants
    None | 0 | 1 | 0 | 1
    Moderate | 1 | 1 | 0 | 2
    Severe | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Most Bothersome Vulvar and Vaginal Atrophy (VVA) Symptom (MBS) of Vaginal Dryness
Description: This outcome measure was analyzed using Cochran-Mantel-Haenszel (CMH) row mean scores test controlling for study center and uterine status. VVA Symptom Score: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe
Time Frame: Baseline (Randomization) to Week 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 102 | 118 | 104
Units on a scale | -1.22 (0.929) | -1.26 (1.025) | -0.84 (0.996)

2. Primary Outcome: Mean Change From Baseline in the MBS of Vaginal Pain Associated With Sexual Activity
Description: This outcome measure was analyzed using CMH row mean scores test controlling for study center and uterine status. VVA Symptom Score: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe
Time Frame: Baseline (Randomization) to Week 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 136 | 120 | 122
Units on a scale | -1.02 (1.132) | -1.19 (1.292) | -0.89 (1.115)

3. Primary Outcome: Mean Change From Baseline in Vaginal pH
Time Frame: Baseline (Screening) to Week 12
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 282 | 276 | 268
pH | -0.67 (1.054) | -1.01 (1.053) | -0.096 (0.8357)

4. Primary Outcome: Mean Change From Baseline in Percentage of Parabasal Cells in Maturation Index of Vaginal Smear
Time Frame: Baseline (Screening) to Week 12
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 280 | 276 | 268
percentage of parabasal cells | -21.9 (32.60) | -30.1 (37.93) | 3.98 (35.205)

5. Secondary Outcome: Change From Baseline in Visual Evaluation of the Vagina
Description: Exam Rating Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe
Time Frame: Baseline (Screening) to Week 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 230 | 223 | 215
Units on a scale
  Petechiae | -0.50 (0.829) | -0.60 (0.848) | -0.037 (0.8080)
  Pallor | -0.75 (0.914) | -0.93 (0.930) | -0.30 (0.940)
  Friability | -0.57 (0.922) | -0.71 (0.911) | -0.16 (0.818)
  Vaginal dryness in mucosa | -1.05 (0.959) | -1.22 (0.981) | -0.48 (0.911)
  Vaginal redness in mucosa | -0.44 (0.811) | -0.60 (0.924) | -0.23 (0.792)

6. Secondary Outcome: Change From Baseline in Severity of VVA Symptoms
Description: as for outcome 2
Time Frame: Baseline (Randomization) to Week 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 282 | 276 | 268
Units on a scale
  Vaginal dryness | -0.96 (1.018) | -1.17 (1.050) | -0.63 (1.047)
  Vaginal pain associated with sexual activity | -0.77 (1.200) | -0.87 (1.278) | -0.57 (1.224)
  Vulvar/vaginal itching or irritation | -0.40 (1.080) | -0.58 (0.982) | -0.44 (0.948)
  Difficult/painful urination | -0.17 (0.676) | -0.20 (0.673) | -0.097 (0.6745)
  Vaginal bleeding associated with sexual activity | -0.26 (0.807) | -0.23 (0.707) | -0.12 (0.667)

7. Secondary Outcome: Change From Baseline in Estradiol Levels
Time Frame: Baseline (Screening) to Week 12
Population: Analysis populations for each hormone:
  Ospemifene(30 mg): E2-231, FSH-232, LH-231, SHBG-232, Testosterone(free)-183, Testosterone(total)-183 Ospemifene(60 mg): E2-221, FSH-222, LH-222, SHBG-221, Testosterone(free)-175, Testosterone(total)-176 Placebo: E2-216, FSH-216, LH-216, SHBG-216, Testosterone(free)-178, Testosterone(total)-178
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 232 | 222 | 216
pg/mL | -1.44 (19.01) | 1.02 (12.74) | 0.30 (3.90)

8. Primary Outcome: Mean Change From Baseline in the Percentage of Superficial Cells in Maturation Index of Vaginal Smear
Time Frame: Baseline (Screening) to Week 12
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 280 | 276 | 268
percentage of superficial cells | 7.78 (12.136) | 10.8 (15.66) | 2.18 (8.393)

9. Secondary Outcome: Change From Baseline in Follicle Stimulating Hormone Levels
Time Frame: Baseline (Screening) to Week 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 232 | 222 | 216
IU/L | -5.93 (12.49) | -8.71 (13.61) | -1.33 (10.87)

10. Secondary Outcome: Change From Baseline in Luteinizing Hormone Levels
Time Frame: Baseline (Screening) to Week 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 232 | 222 | 216
IU/L | -2.85 (6.07) | -3.73 (5.83) | 0.41 (7.25)

11. Secondary Outcome: Change From Baseline in Sex Hormone Binding Globulin Levels
Time Frame: Baseline (Screening) to Week 12
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 232 | 222 | 216
nmol/L | 11.1 (16.46) | 22.8 (22.06) | -2.17 (12.02)

12. Secondary Outcome: Change From Baseline in Testosterone (Free) Levels
Time Frame: Baseline (Screening) to Week 12
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 232 | 222 | 216
ng/dL | 0.002 (0.51) | -0.031 (0.15) | -0.008 (0.13)

13. Secondary Outcome: Change From Baseline in Testosterone (Total) Levels
Time Frame: Baseline (Screening) to Week 12
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 232 | 222 | 216
ng/dL | 1.55 (18.82) | 1.92 (5.56) | -0.059 (6.07)

14. Secondary Outcome: Change From Baseline in Urinary Symptoms
Time Frame: Baseline (Randomization) to Week 12
Measure: Number; unit: Participants
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Number analyzed (Participants) | 229 | 223 | 216
Participants
  Frequent urination-Improved | 49 | 63 | 60
  Frequent urination-Worsened | 24 | 25 | 22
  Urine leakage (feeling of urgency)-Improved | 52 | 53 | 57
  Urine leakage (feeling of urgency)-Worsened | 24 | 26 | 32
  Urine leakage with physical exertion-Improved | 50 | 56 | 47
  Urine leakage with physical exertion-Worsened | 24 | 23 | 27
  Small amount of urine leakage-Improved | 59 | 55 | 58
  Small amount of urine leakage-Worsened | 30 | 32 | 27
  Difficulty emptying bladder-Improved | 25 | 26 | 24
  Difficulty emptying bladder-Worsened | 14 | 11 | 15
  Pain in lower abdominal/genital area-Improved | 37 | 41 | 37
  Pain in lower abdominal or genital area-Worsened | 17 | 13 | 16

ADVERSE EVENTS:
Time Frame: 16 weeks (Visit 2 [Randomization] to Visit 5)
Arm/Group | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant | Placebo Tablets and Nonhormonal Vaginal Lubricant
Serious Adverse Events (participants affected / at risk) | 5/282 | 0/276 | 4/268
Other Adverse Events (participants affected / at risk) | 99/282 | 99/276 | 49/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant (N=282) | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant (N=276) | Placebo Tablets and Nonhormonal Vaginal Lubricant (N=268)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Duodenal Stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Red Blood Cell Sedimentation Rate Increased (Investigations) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Gastric Bypass (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ospemifene 30 mg/Day and Nonhormonal Vaginal Lubricant (N=282) | Ospemifene 60 mg/Day and Nonhormonal Vaginal Lubricant (N=276) | Placebo Tablets and Nonhormonal Vaginal Lubricant (N=268)
Urinary Tract Infection (Infections and infestations) | 20 | 20 | 8
Fungal Infection (Infections and infestations) | 7 | 9 | 1
Sinusitis (Infections and infestations) | 6 | 7 | 10
Vulvovaginal Mycotic Infection (Infections and infestations) | 3 | 11 | 2
Headache (Nervous system disorders) | 17 | 7 | 14
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 | 11 | 4
Vaginal Discharge (Reproductive system and breast disorders) | 12 | 11 | 1
Hot Flush (Vascular disorders) | 27 | 23 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.